CLINICAL TRIAL: NCT02571881
Title: Opioid Induced Bowel Dysfunction in Patients Undergoing Cesarean Section
Acronym: oksisektio
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH01-07-2012
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Constipation; Pain, Postoperative
Keywords: constipation; oxycodone; caesarean section
MeSH Terms: conditions — Constipation; Pain, Postoperative | interventions — Cesarean Section; Oxycodone; oxycodone naloxone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone (Active Comparator): Oxycodone 10 mg prolonged release tablet twice a day after caesarean section
  Interventions: Procedure: Caesarean section; Drug: Oxycodone
- Oxycodone-naloxone (Experimental): Oxycodone-naloxone 10/5 mg prolonged release tablet twice a day after caesarean section
  Interventions: Procedure: Caesarean section; Drug: oxycodone-naloxone

INTERVENTIONS:
Procedure: Caesarean section — After caesarean section oxycodone or oxycodone-naloxone prolonged release tablet twice a day is started for pain medication
Drug: Oxycodone
  Arms: Oxycodone
Drug: oxycodone-naloxone
  Arms: Oxycodone-naloxone

SUMMARY:
Constipation is common in pregnant women. Surgery, anaesthesia and opioid analgesics may further impair bowel function. The aim of the present study was to evaluate if oxycodone-naloxone combination compared to oxycodone reduced bowel dysfunction in patients undergoing caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* • elective caesarean section in spinal anaesthesia

  * normal full term single pregnancy
  * age 18 years or more
  * BMI 20 - 35 kg/m2
  * written informed consent obtained

Exclusion Criteria:

* • not normal or full term pregnancy

  * age less than 18 years
  * allergy to study drugs
  * substance misuse other contraindication to used study drugs no informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with opioid induced bowel dysfunction assessed with bowel function index | time from the first drug intake up to three weeks postoperatively

SECONDARY OUTCOMES:
Oxycodone concentrations in maternal plasma | time before the first drug intake to the day when patient leaves the hospital up to maximum of seven days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Undecided